CLINICAL TRIAL: NCT00396396
Title: Role of Acetylcysteine in Creatinine Clearance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Virginia Medical School (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: EVMS 06-03-FB-0044
Record Dates: First submitted 2006-11-03; First posted 2006-11-06 (Estimated); Last update posted 2006-11-06 (Estimated); Status verified 2006-11

CONDITIONS: Creatinine Clearance
Keywords: Creatinine clearance; Acetylcysteine
MeSH Terms: interventions — Acetylcysteine

INTERVENTIONS:
Drug: Acetylcysteine

SUMMARY:
The purpose of this study is to investigate the exact role of Acetylcysteine (Mucomyst) in altering creatinine clearance. Prior studies have shown the protective effects of Acetylcysteine on contrast-induced renal dysfunction. In these studies, Acetylcysteine lowered the incidence of serum creatinine elevation after administration of radiographic contrast agents. Not only was the increase in serum creatinine prevented, the studies also demonstrated a significant increase in creatinine clearance after administration of the agent. These prior studies did not evaluate if the increase in creatinine clearance was indeed from a protective benefit of Acetylcysteine in preserving the GFR versus simply increasing the proximal tubular creatinine secretion without actually affecting the GFR. We propose an experiment to help support our hypothesis that Acetylcysteine increases creatinine clearance via an increase in proximal tubular secretion of creatinine.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 79 years
2. In good general health
3. Able to provide informed consent

Exclusion Criteria:

1. Allergy to acetylcysteine or cimetidine,
2. Age less than 18 years or greater than 79 years of age,
3. Women of childbearing age and not able to use adequate contraception, or 4. Anyone currently on any medication that interferes with tubular secretion of creatinine such as trimethoprim-sulfamethoxazole (Bactrim).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R McCune, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Eastern Virginia Medical School/Nephrology Associates, Norfolk, Virginia, United States